CLINICAL TRIAL: NCT02350699
Title: Non Blinded Control Study of High School Athletes in Non Contact Sports
Brief Title: Control Study of Nautilus BrainPulse for the Detection of Concussion
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Normal-001
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control: Nautilus BrainPulse
  Interventions: Device: Nautilus BrainPulse

INTERVENTIONS:
Device: Nautilus BrainPulse — A noninvasive device to detect concussion utilizing headset and sensors

SUMMARY:
To use the Nautilus BrainPulse to compare and contrast the signal patterns from this cohort's signal patterns with those of concussed high school athletes.

DETAILED DESCRIPTION:
This study is a non-blinded study in high school athletes who will be presumed to no be suffering from a concussion. Healthy controls will be recruited from high school sports that are not associated with physical contact, which could generate concussions.

The primary objective of this study is to improve Jan Medical's signal analysis. Jan Medical will perform analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 14 and 19 years of age
* Participating in non-contact sport at the Freshman, JV, and varsity level in a Bay Area High School
* Able to provide signed informed consent or have a legally authorized representative willing to provide informed consent on the subject's behalf

Exclusion Criteria:

* History, if any, of concussion or stroke
* History, if any, of alcohol or drug abuse
* History, if any, of mental disorder or cerebrovascular disorder
* Pregnant women
* Failure to comply with recording schedule
* Not suitable for participation in the study in the opinion of the PI
* Have suffered a concussion during the study
* Plays a contact sport (ex- football, lacrosse, basketball, soccer, ice hockey, cross-country)
* Related to a Jan Medical employee

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects who are healthy controls and participate in a non-contact sport at the high school level.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To collect non-blinded Nautilus BrainPulseTM recordings from high school athletes who do not participate in a contact sport | 4 months
  BrainPulse recordings collected in this study will be used as an age-matched control cohort for comparison with already collected concussion data that is under development for identifying a concussion algorithm. The device recordings will be visually compared for similarities and differences using data mining practices looking for features that are consistent between the concussion subjects and healthy normals.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lovoi, PhD, Principal Investigator — Jan Medical, Inc.
Locations (1):
- Jan Medical, Inc., Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No